CLINICAL TRIAL: NCT00318084
Title: The Proton Pump Inhibitor Test in Reflux Disease: a Study Using Nexium in General Practice Patients
Brief Title: PPI Test in GP Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: UMC Utrecht (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25N54
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: GERD
Keywords: Gastroesophageal reflux disease; Heartburn; Acid-related diseases; Acid reflux disease; Nexium
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole; Ambulatory Care Facilities

INTERVENTIONS:
Drug: Esomeprazole
Procedure: Ambulatory 24-hour esophageal pH-monitoring

SUMMARY:
The purpose of this study is to determine the diagnostic value of two week treatment with Nexium as a confirmatory test for patients with suspected reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptoms suggestive for gastric acid reflux disease during 2 or more days per week

Exclusion Criteria:

* Treatment with prokinetic or acid secretion inhibitors within 4 weeks prior to inclusion
* Treatment with a PPI for more than 30 days within the last 3 months prior to inclusion
* History of proven peptic ulcer disease, unless successfully treated with Helicobacter pylori eradication longer than 1 month before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01

PRIMARY OUTCOMES:
Diagnostic test characteristics and the positive and negative predictive value of a 2-week Nexium-based PPI test using symptom analysis of 24-hour esophageal pH monitoring as gold standard.

SECONDARY OUTCOMES:
To assess the optimal duration of a Nexium-based PPI test, and the predictive value of different symptoms for presence of reflux-related symptoms.
Obtain information on patient satisfaction, the course of reflux symptoms, the consumption of acid suppressing drugs, the disease-related quality of life at a follow up periods of 3 months in patients with a positive and negative PPI test.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, Study Director — AstraZeneca
Locations (1):
- Research Site, Utrecht, Netherlands